CLINICAL TRIAL: NCT01539278
Title: Effect of Adenotonsillectomy on Quality of Life in Children With Mild Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Children's Hospital of The King's Daughters (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-12-FB-0266
Record Dates: First submitted 2012-02-16; First posted 2012-02-27 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea, Obstructive; Child; Tonsillectomy; Adenoidectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation, no surgery (control) (Active Comparator): Patients have been diagnosed with mild OSA, no intervention is done; enrolled patients may be randomly or nonrandomly placed in this group
  Interventions: Other: Observation alone / no intervention
- Surgery (adenotonsillectomy) (Experimental): Patients who have been diagnosed with mild OSA. Patient may be randomly assigned or non-randomly choose to be in this group; all undergo adenotonsillectomy
  Interventions: Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: Adenotonsillectomy — Tonsils and adenoids are surgically removed
  Other Names: T&A
  Arms: Surgery (adenotonsillectomy)
Other: Observation alone / no intervention — Patients are observed over time, no surgery is done, subjects complete QOL questionnaires at set intervals
  Arms: Observation, no surgery (control)

SUMMARY:
In children, enlarged adenoids and/or tonsils are the most common cause of obstructive sleep apnea (OSA), which is temporary blockage of breathing during sleep. Surgery to remove the tonsils and adenoids is the first-line treatment for disorder, and has been shown to cure the majority of children. However, for children with only a mild degree of OSA and few symptoms, surgery is less clear-cut, since two-thirds of these children do not develop worsening disease.

Research shows that some children with mild OSA and behavior problems are helped by removing the tonsils and adenoids. In children with all degrees of OSA, surgery has improved scores on tests that measure quality of life (QOL).

The investigators hypothesize that children with mild OSA will demonstrate changes on QOL assessment following adenotonsillectomy. These findings may help to guide the surgeon in selecting the children with mild OSA who are more likely to benefit from surgery.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a sleep-related breathing disorder that is characterized by intermittent episodes of upper airway collapse and cessation of airflow during sleep. It comprises the severest extent of a spectrum of sleep disordered breathing (SDB) which includes primary snoring and upper airway resistance syndrome. OSA is a cause cardiovascular morbidity in adults and children and a public health concern, affecting 2-4% of the middle aged population (Giles 2009) and 2-3% of children in the United States (Katz 2010). It is further associated with an increased mortality risk in adults (Giles 2009) and well-described metabolic, cardiovascular, and neuropsychological deficits in children (Katz 2010). The latter symptoms include changes in behavior, memory and cognition, and poor school performance.

In children, adenotonsillar hyperplasia is uniformly the most common cause of upper airway obstruction, and the first-line therapy for these children is adenotonsillectomy (Darrow 2007). While its effectiveness is complicated by children with obesity and other comorbidities, the most recent analyses of outcomes using postsurgical apnea-hypopnea index reveal that adenotonsillectomy alone is able to cure approximately 60% of child OSA (Friedman 2010). Improvements have also been shown with neuropsychological outcomes such as behavior, school performance, attention, and others. (Katz 2010).

"Mild OSA" is an evolving definition; it is characterized by the polysomnographic finding of AHI range greater than 1 and less than 5, defined by Katz and Marcus.(Wagner 2007) This range corresponds to the difference in the defined pathological minimum AHI for children (normal AHI < 1) and adults (normal AHI < 5). In practice, "mild OSA" remains a common reason for delaying adenotonsillectomy in an otherwise asymptomatic child, since children with mild OSA have been shown to exhibit neurocognitive functioning equivalent to controls.(Calhoun 2009) However, psychosocially these children often have problems, and adenotonsillectomy has been shown to improve these children's behavior as measured by atypicality, depression, hyperactivity, and somatization.(Mitchell 2007) Furthermore, among one-third of children with mild OSA, the natural history is progression of disease.(Li 2010)

Psychosocial problems also become manifest using health-related quality-of-life (QOL) symptom scores. The study of QOL in children with OSA has become an area of scholarly interest in the last 15 years. It was only in 2000 that an OSA-specific QOL questionnaire was first developed and validated for use in children (2000 Franco). A recent meta-analysis of QOL following adenotonsillectomy revealed significant improvements in QOL scores in patients undergoing surgery for all severity levels of OSA.(2008 Baldassari) This meta-analysis included studies using validated QOL instruments, namely the Child Health Questionnaire (CHQ) and OSA-18.

Only one study of QOL in children with mild OSA found no clinically significant differences between patients who underwent adenotonsillectomy and controls; however, disease-specific QOL instrument (such as the OSA-18) was not used.(van Staaij 2004)

The investigators hypothesize that children with mild OSA will demonstrate changes on QOL assessment following adenotonsillectomy, particularly in OSA-specific domains. If true, a threshold for preoperative QOL scores may serve as a relative indication for adenotonsillectomy in the setting of mild OSA, independent of behavioral issues.

ELIGIBILITY:
Inclusion Criteria:

* Any obstructive breathing symptoms such as snoring, mouth-breathing, sleep pauses, gasping, restless sleep, witnessed apneas, daytime somnolence, and enuresis.
* Children between the ages of 3-16 years of age that have had a sleep study with an Apnea Hypopnea Index (AHI) score of 1 to 5.

Exclusion Criteria:

* Subject/LAR unwillingness to comply with all study procedures
* Prior otolaryngologic surgery
* Prior sleep study
* Pregnant or breastfeeding
* Under 3 years of age and older than 16 years of age
* Congenital head and neck malformations or other syndromes

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Health-related Quality of Life (HR-QOL) from baseline, as measured by the OSA-18 Questionnaire and Children's Health Questionnaire (CHQ-28) | baseline, 3 months, 6 months
  HR-QOL forms OSA-18 and CHQ-28 to be completed by subjects at the time of enrollment, and at thereafter at three and six months. Main outcome measure is the difference or change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M. Baldassari, MD, Principal Investigator — Eastern Virginia Medical School Dept. of Otolaryngology-Head & Neck Surgery; Children's Hospital of the King's Daughters
Locations (1):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States

REFERENCES:
- [Background] Baldassari CM, Mitchell RB, Schubert C, Rudnick EF. Pediatric obstructive sleep apnea and quality of life: a meta-analysis. Otolaryngol Head Neck Surg. 2008 Mar;138(3):265-273. doi: 10.1016/j.otohns.2007.11.003. PMID 18312869
- [Background] Calhoun SL, Mayes SD, Vgontzas AN, Tsaoussoglou M, Shifflett LJ, Bixler EO. No relationship between neurocognitive functioning and mild sleep disordered breathing in a community sample of children. J Clin Sleep Med. 2009 Jun 15;5(3):228-34. PMID 19960643
- [Background] Darrow DH. Surgery for pediatric sleep apnea. Otolaryngol Clin North Am. 2007 Aug;40(4):855-75. doi: 10.1016/j.otc.2007.04.008. PMID 17606027
- [Background] Friedman M, Wilson M, Lin HC, Chang HW. Updated systematic review of tonsillectomy and adenoidectomy for treatment of pediatric obstructive sleep apnea/hypopnea syndrome. Otolaryngol Head Neck Surg. 2009 Jun;140(6):800-8. doi: 10.1016/j.otohns.2009.01.043. PMID 19467393
- [Background] Giles TL, Lasserson TJ, Smith BH, White J, Wright J, Cates CJ. Continuous positive airways pressure for obstructive sleep apnoea in adults. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD001106. doi: 10.1002/14651858.CD001106.pub3. PMID 16855960
- [Background] Gozal D. Sleep, sleep disorders and inflammation in children. Sleep Med. 2009 Sep;10 Suppl 1:S12-6. doi: 10.1016/j.sleep.2009.07.003. Epub 2009 Jul 31. PMID 19647481
- [Background] Katz ES, D'Ambrosio CM. Pediatric obstructive sleep apnea syndrome. Clin Chest Med. 2010 Jun;31(2):221-34. doi: 10.1016/j.ccm.2010.02.002. PMID 20488283
- [Background] Li AM, Au CT, Ng SK, Abdullah VJ, Ho C, Fok TF, Ng PC, Wing YK. Natural history and predictors for progression of mild childhood obstructive sleep apnoea. Thorax. 2010 Jan;65(1):27-31. doi: 10.1136/thx.2009.120220. Epub 2009 Sep 23. PMID 19776090
- [Background] Mitchell RB, Kelly J. Behavioral changes in children with mild sleep-disordered breathing or obstructive sleep apnea after adenotonsillectomy. Laryngoscope. 2007 Sep;117(9):1685-8. doi: 10.1097/MLG.0b013e318093edd7. PMID 17667138
- [Background] van Staaji BK, van den Akker EH, Rovers MM, Hordijk GJ, Hoes AW, Schilder AG. Effectiveness of adenotonsillectomy in children with mild symptoms of throat infections or adenotonsillar hypertrophy: open, randomised controlled trial. Clin Otolaryngol. 2005 Feb;30(1):60-3. doi: 10.1111/j.1365-2273.2005.00980.x. PMID 15748193
- [Background] Wagner MH, Torrez DM. Interpretation of the polysomnogram in children. Otolaryngol Clin North Am. 2007 Aug;40(4):745-59. doi: 10.1016/j.otc.2007.04.004. PMID 17606021